CLINICAL TRIAL: NCT06220903
Title: The Effect of Complex Decongestive Therapy on Fluid Excretion From The Body in Patients With Lymphedema
Brief Title: The Effect of Complex Decongestive Therapy in Patients With Lymphedema
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Dilanur Özkaraoğlu, PT, MSc, Assistant Professor, Medipol University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MedipolU-FTR-DO-02
Record Dates: First submitted 2024-01-15; First posted 2024-01-24 (Actual); Last update posted 2024-01-25 (Actual); Status verified 2024-01

CONDITIONS: Lymphedema; Urine Marking; Quality of Life; Edema
MeSH Terms: conditions — Lymphedema; Edema

STUDY DESIGN:
Intervention Model Description: A study group that received treatment and was monitored for a total of 20 sessions every day.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment Group (Experimental): Complex DecongestivePhysiotherapy program was planned for the affected extremity of the cases. The treatment was performed 5 days a week, for 4 weeks, for a total of 20 sessions and each session was 60 minutes. The treatment included Manual Lymph Drainage, skin care, multi-layer bandaging, exercise and compression stockings.
  Interventions: Other: Complex Decongestive Therapy

INTERVENTIONS:
Other: Complex Decongestive Therapy — 1. Manual Lymph Drainage: Cervical region lymph drainage and abdominal region lymph drainage (especially combined with abdominal breathing) were applied.
  2. Skin Care: Moisturizing creams with a pH of 5.5 were applied to the extremities before bandaging.
  3. Multilayer Bandaging: Short pull bandage application was applied in a gradient manner.
  4. Exercise: Joint range of motion exercises, breathing exercises (abdominal breathing), decongestive exercises, and self-drainage techniques were taught.
  5. Compression Stocking: After the decongestion phase was over, flat knit compression stockings were recommended according to the patient's extremity.

SUMMARY:
The aim of this study is to investigate objectively the effect of lymphatic fluid which is circulated with Complex Decongestive Therapy on fluid excretion from the body in patients with lymphedema.

DETAILED DESCRIPTION:
The lymphatic system is the accessory circulatory system that takes lymph fluid from the interstitial space and adds it to the blood circulation. It starts from the interstitial space. It consists of lymph vessels, lymph fluid and lymphatic organs. Lymph fluid passes through many lymph nodes during its transport and is filtered in these nodules. The lymphatic system takes lymphatic fluid from the tissues and brings it to the venous part of the circulatory system. The main task of the lymph system is to reabsorb substances that cannot be absorbed by the blood circulation system. Non-absorbable substances in the interstitial space are called lymphatic load. Lymphatic load; It consists of protein, water, fat and cells. The aim of lymphedema treatment is to remove the protein-rich fluid accumulated in the interstitial space into the venous system. There are many factors in the flow of lymph fluid into the veins. The most important of these is the high filtration pressure that occurs when fluid is filtered through blood capillaries. Lymph fluid flowing from the periphery to the center is generally affected by pressure changes and moves from where the pressure is high to where it is low. Contraction of the muscles adjacent to the lymph vessels, pulsation of the neighboring arteries, and the effect of the smooth muscles in the lymph vessel wall also cause pressure changes. Other factors include respiratory movements acting as a pump in the lymph flow, the actual pressure effect of abdominal pressure on the cisterna chyli, and negative intrathoracic pressure.

Complex Decongestive Physiotherapy is proven effective and considered the gold standard for the treatment of lymphedema. It increases the hydrostatic pressure that has decreased due to edema and helps the lymph fluid to re-enter the circulation.

Purpose of the study; To objectively investigate whether the lymph fluid added to the circulation through Complex Decongestive Physiotherapy in lymphedema patients has an effect on fluid excretion from the body.

ELIGIBILITY:
Inclusion Criteria:

* Female cases
* Cases diagnosed with lower extremity unilateral/bilateral lymphedema
* Having received or not received radiotherapy and/or chemotherapy

Exclusion Criteria:

* Having received treatment for lymphedema in the last year
* Having metastatic disease
* Those diagnosed with severe heart failure and/or arrhythmia
* Arterial disorders
* Kidney diseases
* Infection in affected extremities
* Psychological disorders
* Diabetes
* Nephrotic syndrome
* Diuretic use
* Patients using chemotherapy and drugs that have toxic effects on the kidneys
* Those with liver cirrhosis, liver disease
* Neurological diseases

Ages: 30 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
MoistureMeterD Compact Device | 4 weeks
  Tissue dielectric constant technique provides information about the emergence of lymphedema in the early stages and the change in the amount of water under the skin. A high-frequency electromagnetic wave produced by the device is directed to the skin by contacting the probe with the skin. The effective measurement depth is 2.5 mm. The device evaluates the amount of water under the tissue thought to be the beginning of lymphedema.
Liquid Intake-Urine Excretion Tracking | 4 weeks
  The subjects were asked to fill out a 24-hour fluid intake-urine excretion chart to evaluate the difference between fluid intake and urine excretion.

SECONDARY OUTCOMES:
Body Mass Index | 4 weeks
  BMI values of the cases; Calculated and recorded using TANITA MC 780 S Professional Body Analysis Monitor. It was calculated with the formula Body Mass Index (BMI) = Weight/Height2 (kg/m2).
Range of motion | 4 weeks
  Universal Goniometer was used to evaluate joint range of motion. Hip, knee and foot flexion were measured.
Evaluation of edema | 4 weeks
  While the patients were in a semi-sitting position and the foot and ankle were in neutral position, circumference measurements were made with a tape measure at 5 cm intervals from the ankle to the lateral malleolus level towards the proximal. Extremity volume was determined by calculating with the frustum formula. The difference between both extremities (healthy and diseased side) was determined and measurements were made every day before and during treatment.
Lymphedema Quality of Life | 4 weeks
  The patients' quality of life was evaluated using the Lymphedema Quality of Life Questionnaire-Lower extremity, which consists of questions about symptoms, body image, function and mode, respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Cemile Uydur, MsC, Principal Investigator — Avrupa Şafak Hospital Physical Therapy and Rehabilitation Unit
Locations (1):
- Istanbul Medipol University, Istanbul, Beykoz, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No